CLINICAL TRIAL: NCT04805047
Title: Sodium Restriction by Behavioral Intervention: Education and Monitoring
Brief Title: SodiUm Restriction by Behavioral Intervention
Acronym: SURBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: XJTU1AF2020LSK-073
Record Dates: First submitted 2021-03-17; First posted 2021-03-18 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention:education and monitoring (Experimental): regular education programs supported by a dietician in combination with urine sodium monitoring as a feedback
  Interventions: Behavioral: education and monitoring
- control (No Intervention): regular care

INTERVENTIONS:
Behavioral: education and monitoring — regular education programs supported by a dietician in combination with urine sodium monitoring as a feedback
  Arms: Intervention:education and monitoring

SUMMARY:
The aim of this study is to evaluate the effects and efficacy of dietary sodium restriction by mean of a new healthcare approach in patients with immunoglobulin A nephropathy. The test persons in the intervention group are actively supported to adhere to a restricted sodium diet with a structured education program in combination with regular sodium excretion monitoring.

DETAILED DESCRIPTION:
Patients in the intervention group receive regular sodium-restriction education by a dietician, which entails introducing food types and cooking skills, quantifying salt intake with a special spoon and recording detailed interactive food diary. Sodium excretion was measured using one 24-hour urine collection regularly to assess dietary compliance and enable feedback. The test persons with sodium excretion higher than 90mmol/24h will receive intensive education. Test persons in the control group receive standard care. After 2 weeks in study, all test persons visit the outpatient clinic for measurements and data collection. Within 3 months of total study duration, data collection and measurements take place at the end of every month.

At each timepoint blood and 24-hourly urine is collected, test persons fill out questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients>14 years of age and <70 years of age
* Diagnosed immunoglobulin A nephropathy with biopsy;
* eGFR>30ml/min per 1.73m2 using Chronic Kidney Disease Epidemiology Collaboration formula
* Proteinuria >1 g per day
* urinary sodium excretion >200 mmol per day within one month
* systolic blood pressure higher than 140 mmHg or diastolic blood pressure higher than 90 mmHg, or a well-controlled blood pressure by treatment with antihypertensives including renin-angiotensin-aldosterone system-blockade (ACE-inhibitor or ARB)
* Written informed consent

Exclusion Criteria:

* Be treated with diuretics
* Blood pressure > 180 mmHg systolic or > 125 mmHg diastolic without medical treatment
* Have undergone renal transplantation
* With acute kidney injury (RIFLE criteria) < 6 months ago
* Cardiovascular or cerebrovascular event (myocardial infarction, cerebral hemorrhage or infarction) < 6 months ago
* With progressive malignancy or pregnancy
* With contraindications of RAAS blockers
* unwilling or unable to meet the requirements of the protocol

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
24 hour urine protein excretion | 3 months
  24 hour urine protein excretion after 3 months

SECONDARY OUTCOMES:
24 hour urine sodium excretion | 3 months
  24 hour urine sodium excretion after 3 months
blood pressure | 3 months
  blood pressure after 3 months
estimated Glomerular Filtration Rate change | 3 months
  estimated Glomerular Filtration Rate change after 3 months
Psychological well-being | 3months
  Psychological well-being will be assessed with multiple choice questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Huixian Li, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First affiliated hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639